CLINICAL TRIAL: NCT06946849
Title: Second-line Regimen Combined With Radiotherapy Versus Without Radiotherapy in Patients With Locally Advanced/Oligometastatic Intrahepatic Cholangiocarcinoma After Failure of First-line Treatment：an Open-label, Randomized, Controlled Phase II Clinical Study
Brief Title: Second-line Regimen Combined With Radiotherapy Versus Without Radiotherapy in Patients With Locally Advanced/Oligometastatic ICC After Failure of First-line Treatment：an Open-label, Randomized, Controlled Phase II Clinical Study
Acronym: SED-RO-ICC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Zeng Zhaochong, professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025087; KY2025XXX (Registry Identifier: Zhongshan Hospital, Fudan University)
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc)
Keywords: Intrahepatic Cholangiocarcinoma, Radiotherapy, Second-line regimen
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension | interventions — Radiotherapy; Folfox protocol; regorafenib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2L SoC+RT (Experimental): 2L SoC regimen combined with radiotherapy
  Interventions: Radiation: radiotherapy; Drug: FOLFIRI or FOLFOX or Regorafenib
- 2L-SoC (Active Comparator)
  Interventions: Drug: FOLFIRI or FOLFOX or Regorafenib

INTERVENTIONS:
Radiation: radiotherapy — Radiotherapy
  Arms: 2L SoC+RT
Drug: FOLFIRI or FOLFOX or Regorafenib — FOLFIRI or FOLFOX or Regorafenib

SUMMARY:
Second-line regimen with or without consolidative radiotherapy in patients with oligometastatic/locally advanced unresectable intrahepatic cholangiocarcinoma: an open-label, randomised, controlled study.

DETAILED DESCRIPTION:
Second-line regimen with or without consolidative radiotherapy in patients with oligometastatic/locally advanced unresectable intrahepatic cholangiocarcinoma: an open-label, randomised, controlled study. Eligible patients will be randomized in a 1:1 ratio to receive either second-line regimen alone (control arm) or second-line regimen plus consolidative radiotherapy to all sites of known disease (investigational arm). patients in both arms have the option of receiving upfront or subsequent standard palliative radiotherapy to any symptomatic sites requiring prompt intervention. Because of the different treatment modalities in the study, it is not possible to blind the patient or physician to the treatment arm. Follow-up for tumor assessment will conclude 52 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* (1) Advanced or metastatic intrahepatic cholangiocarcinoma confirmed by histopathology that cannot be surgically removed.

  (2) Failed to receive first-line standard treatment. (3) Definition of oligometastatic/locally advanced unresectable BTC disease: not a candidate for surgical resection at all sites: surgery to all sites not recommended by multidisciplinary team, or unfit or declining surgery.

  (4) Definition of oligometastatic disease: patients with distant organ metastasis or nonregional lymph node metastasis, or distant organ/nonregional lymph node metastasis and regional lymph node metastasis, as defined by the American Joint Committee on Cancer, 8th edition. The total number of metastases is ≤5 and the number of metastases in any single organ system (e.g., lung, liver) is ≤3.

  (4) All sites of disease must be amenable to radiotherapy and can be safely treated. Each lesion is counted separately at the time of registration and contributes to the total number of metastases. For regional lymph nodes metastases, all positive regional lymph nodes are counted together as one lesion. For nonregional lymph node metastases, adjacent metastatic lymph nodes can be treated as one lesion. Lesions that have subsided during previous treatment (i.e., are no longer visible on CT scan or have eliminated affinity on positron emission tomography [PET]-CT) are not included in the total number. At least one metastatic lesion meets the RECIST v1.1 criteria for assessable lesions. Bone metastases without soft tissue involvement can be included but are not considered assessable lesions. However, if bone metastases have soft tissue involvement and meet the criteria for assessable lesions, they are considered measurable lesions.

  (5) Patients who experience recurrence after curative surgery with a time interval of >6 months can be eligible for inclusion. If adjuvant therapy (excluding radiotherapy) is administered, the patient must have completed adjuvant therapy for a period of at least 6 months before meeting the inclusion criteria.

  (5) Primary tumor lesions and all metastases of current diagnosis have not received local treatment, such as radiotherapy, surgery or radiofrequency ablation, prior to enrollment.

  (6) The patient is over 18 years old and has an Eastern Cooperative Oncology Group score of 0-1; (7) Life expectancy is greater than 12 weeks. (8) Vital organ function meets the following requirements: absolute neutrophil count ≥1.5 × 109/l; platelet count ≥100 × 109/l; hemoglobin ≥9 g/dl; serum albumin ≥2.8 g/dl; total bilirubin ≤1.5 × upper limit of normal (ULN) and alanine transaminase, aspartate aminotransferase and/or alkaline phosphatase ≤2.5 × ULN (if there is liver metastasis, alanine transaminase and/or aspartate aminotransferase ≤5 × ULN; if there is liver metastasis or bone metastasis, alkaline phosphatase ≤5 × ULN); serum creatinine ≤1.5 × ULN or creatinine clearance >60 ml/min. For patients with pulmonary lesions or previous lung irradiation who are known or suspected to have impaired lung function, the forced expiratory volume for 1 second of lung function must be above 1 l.

  (9) Female subjects of childbearing age must have a negative urine or serum pregnancy test within 72 h prior to randomization. Subjects must agree to adequate contraception during the trial.

  (10) Each patient is voluntarily enrolled, and the informed consent form is signed by the patient or their legal representative.

Exclusion Criteria:

* (1) Histology includes components of mixed hepatocellular carcinoma, fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, or biliary adenocarcinoma.

  (2) Complete response to four cycles of first-line systemic treatment (i.e. no measurable target for radiotherapy).

  (3) There is new metastasis during the four cycles of first-line systemic treatment and the number of metastases is more than five.

  (4) Patient has uncontrolled brain metastases or vertebral body metastasis with spinal cord compression symptoms.

  (5) The toxicity of previous antitumor treatment has not recovered to ≤1 based on National Cancer Institute Common Terminology Criteria for Adverse Events v4.03 (except for hair loss) or the level specified by the inclusion/exclusion criteria.

  (6) Patient has uncontrolled pleural, pericardial or pelvic effusion that requires repeated drainage.

  (7) Patient is a pregnant or breastfeeding woman. (8) Patient has a history of immunodeficiency or severe medical disease that is not well controlled and may have an effect on study treatment.

  (9) Any other malignant tumor has been diagnosed within 5 years prior to or after the diagnosis of BTC, except for malignant tumors with a low risk of metastasis and death (5-year survival rate >90%), such as well-treated basal cell or squamous cell skin cancer or cervical cancer in situ.

  (10) Any other condition which in the judgment of the investigator would make the patient inappropriate for entry into this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 2 years
  PFS is will be measured from the randomization to progression or death from any cause. Progression includes enlargement of target lesions and development of new distant metastases and will be assessed using RECIST 1.1.

SECONDARY OUTCOMES:
OS | Up to 2 years
  OS will be the time from randomization until death from any cause.
LCR | Up to 2 years
  Local control of all metastases (refers to all lesions present at time of randomization) will be measured from date of randomization until progression of target lesions.
AEs | Up to 2 years
  Toxicity will involve treatment-related toxicity, including early and late toxicity, as assessed using Common Terminology Criteria for Adverse Events v5.0. All adverse events occurring from randomization until 3 months after the end of treatment, regardless of relatedness to study medication, will be recorded as acute toxicities. Adverse events considered relevant and occurring later than 3 months after the end of treatment will be recorded as late toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaochong Zeng, Principal Investigator — Zhongshan Hospital, Fudan Unuversity; Guoming Shi, Principal Investigator — Zhongshan Hospital, Fudan Unuversity
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No